CLINICAL TRIAL: NCT02242305
Title: A Randomized, Double-blind, Double-dummy, Active-controlled, Parallel-group, Multi-center Trial, in Contrast With Hyoscine Butylbromide Capsule 10mg, to Evaluate the Efficacy and Safety of Hyoscine Butylbromide Tablets 10 mg (20mg, 3 Times Daily, Orally) Over a Period of 3 Days for the Treatment of Occasional or Recurrent Episodes of Self-reported Gastric or Intestinal Spasm-like Pain
Brief Title: Study to Evaluate the Efficacy and Safety of Hyoscine Butylbromide Tablets for the Treatment of Occasional or Recurrent Episodes of Gastric or Intestinal Spasm-like Pain or Discomfort
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202.838
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Hyoscine Butylbromide - Tablet (Experimental)
  Interventions: Drug: Hyoscine Butylbromide - Tablet; Drug: Placebo
- Hyoscine Butylbromide - Capsule (Active Comparator)
  Interventions: Drug: Hyoscine Butylbromide - Capsule; Drug: Placebo

INTERVENTIONS:
Drug: Hyoscine Butylbromide - Tablet
  Arms: Hyoscine Butylbromide - Tablet
Drug: Hyoscine Butylbromide - Capsule
  Arms: Hyoscine Butylbromide - Capsule
Drug: Placebo

SUMMARY:
In contrast with Hyoscine Butylbromide Capsule 10mg, Study is to evaluate the efficacy and safety of Hyoscine Butylbromide tablets 10 mg (20mg, 3 times daily, orally) over a period of 3 days for the treatment of occasional or recurrent episodes of self-reported gastric or intestinal spasm-like pain or discomfort

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent given by the patient
2. Male and female patients aging from 18 to 70
3. Subjects with occasional or recurrent episodes of gastric or intestinal spasm-like pain, or discomfort, such as occur e.g. in irritable bowel syndrome, which has been present for at least 3 months
4. The pain intensity score upon screening is at least 4 cm in VAS score

Exclusion Criteria:

1. Patients with the following concomitant disease were not eligible for enrolment

   * Painful gastric or intestinal spasm of organic origin such as Crohn's disease, ulcerative colitis, lactose intolerance, gastritis, ulcer. Exception: diverticulitis and mild gastritis if dominant symptom was cramp pain, but ineligible if heartburn or reflux were dominant symptoms
   * Pain related with malignancy
   * Patients with other severe pain states of organic origin
   * Mechanical stenosis of the gastrointestinal tract, megacolon
   * Urinary retention associated with mechanical stenosis of urinary tract
   * Narrow-angled glaucoma
   * Tachyarrhythmia
   * Myasthenia gravis
   * Meulengracht-Gilbert syndrome
   * Known depression or known mental illness, anxiety disturbance
2. Frequent vomiting that might have prevented adequate absorption of the active ingredient after the film-coated tablet was taken
3. Patients taking the following concomitant medication are not eligible for enrolment

   * Analgesics
   * Spasmolytics
   * Anticholinergics
   * Affecting gastrointestinal motility, such as propantheline metoclopramide, cisapride, loperamide, diphenoxylate, opioid analgesics, antacids and other ulcer treatment
   * Regular administration of laxatives
   * Narcotics
   * Antidepressant treatment or treatment with psychoactive drugs
4. Pregnancy and/or lactation or planned pregnancy
5. Known hypersensitivity to N-butylscopolammonium bromide
6. Alcohol or drug abuse
7. Simultaneous participating in another clinical trial, or discontinuing from another clinical trial before randomization (administration of study medication); moreover, in the case of screening failure or premature discontinuing from the trial, repeated enrolment is forbidden
8. Unwilling to or unable to complete the entire trial procedure according to the protocol
9. In investigator's opinion, the patient was not proper for the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2009-07-20 (Actual); Study Completion 2009-07-20 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Hyoscine Butylbromide - Tablet (Tab.): The subjects administered Hyoscine Butylbromide (10 mg), (Brand name: Buscopan) sugar coated tablet 20 mg orally, 3 times daily for 3 days.
- Hyoscine Butylbromide - Capsule (Cap.): The subjects administered Hyoscine Butylbromide (10 mg), (Brand name: Jie Jing Ning) sugar coated capsule 20 mg orally, 3 times daily for 3 days.
Period: Overall Study
Arm/Group | Hyoscine Butylbromide - Tablet (Tab.) | Hyoscine Butylbromide - Capsule (Cap.)
Started | 151 | 151
Completed | 145 | 141
Not Completed | 6 | 10
Not completed — Without spasm-like pain during 3 weeks | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance dosing regimen or visit | 2 | 2
Not completed — Subject withdraws inform consent | 0 | 4
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): According to the Intent-to-Treat (ITT) principle, all randomized subjects who took at least one dose of study medication and who provided any data for the primary efficacy endpoint were used in FAS.
  Baseline participants less than participant flow as no abdominal pain within 3 weeks following randomization were withdrawn.
Groups:
- Hyoscine Butylbromide - Tablet: The subjects administered Hyoscine Butylbromide (10 mg), (Brand name: Buscopan) sugar coated tablet 20 mg orally, 3 times daily for 3 days.
- Hyoscine Butylbromide - Capsule: The subjects administered Hyoscine Butylbromide (10 mg), (Brand name: Jie Jing Ning) sugar coated capsule 20 mg orally, 3 times daily for 3 days.
- Total: Total of all reporting groups
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule | Total
Number analyzed (Participants) | 146 | 142 | 288
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (12.49) | 41.9 (12.05) | 42.6 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 84 | 173
  Male | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: Change of the Mean Pain Intensity Score Measured on a Visual Analogue Scale (VAS) Within 3 Days (and Within 1 Day) - ANCOVA
Description: The endpoint presents change of the mean Visual Analogue Scale (VAS) of pain intensity score, recorded daily by the patient in the evening in his/her patient diary describing pain intensity during the previous 24 hours, from the baseline pain intensity. The baseline pain intensity was the pain intensity of first episode on Day 1 after randomization before taking study medication. The mean VAS pain intensity score was calculated for the 3-day treatment period. A VAS for describing the pain intensity was used (VAS: maximum score of 10 cm, the score from 0 - 10 cm reaching from "no pain" to "the most severe pain imaginable").
Time Frame: 3 days (1 day)
Population: Per-Protocol Set (PPS): All randomized subjects in FAS without any major protocol violation were included into the per protocol set, including those subjects who had good treatment compliance (80% to 120%), who did not take any restriction medications during the study period and whose Case Report Form (CRF) was complete as requested.
Measure: Number; unit: Units on a scale
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Number analyzed (Participants) | 141 | 140
Units on a scale
  Within 3 days | -2.48 (1.968) | -2.45 (1.879)
  Within 1 day | -2.36 (1.984) | -2.31 (1.914)
Statistical Analysis 1: Comparison: Hyoscine Butylbromide - Tablet vs Hyoscine Butylbromide - Capsule; Test type: Superiority or Other; p = 0.809, ANCOVA; Analysis of Covariance (ANCOVA) model including treatment and center as fixed effects and baseline pain intensity as a covariate was used; Mean Difference (Final Values) = -0.03, 90% CI 2-sided [-0.33 to 0.27] — Treatment differences were estimated by reference to the Least Squares (LS) mean differences within 3 days and the corresponding 90% CIs. The mean difference calculated as Hyoscine Butylbromide tablets 10 mg - Hyoscine Butylbromide capsules 10 mg
Statistical Analysis 2: Comparison: Hyoscine Butylbromide - Tablet vs Hyoscine Butylbromide - Capsule; Test type: Superiority or Other; p = 0.809, ANCOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.05, 95% CI 2-sided [-0.39 to 0.33] — Treatment differences were estimated by reference to the Least Squares (LS) mean differences within 1 day and the corresponding 90% CIs. The mean difference calculated as Hyoscine Butylbromide tablets 10 mg - Hyoscine Butylbromide capsules 10 mg

2. Secondary Outcome: Change of the Pain Frequency Assessed on 4-stage Verbal Rating Scale (VRS)
Description: The endpoint presents frequency improvement, change of the pain frequency from baseline pain frequency for each of Day 1 - 3. Baseline pain frequency meant the pain frequency before randomization on visit 1. VRS score of Day 3 change from baseline was calculated. A retrospective assessment was entered by the patient in the patient diary, again once daily in the evening, of the pain frequency over the preceding 24 hour period. This was based on a 4-stage Verbal Rating Scale (VRS) with the following scores to the question: "How many times have the spasm-like pains occurred today?" 0 = not at all, 1 = 1-2 times, 2 = 3-5 times, 3 = more than 5 times.
Time Frame: Up to 3 days.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Number analyzed (Participants) | 141 | 140
Units on a scale
  Day 1-Baseline | -0.4 (0.77) | -0.2 (0.73)
  Day 3-Baseline | -1.0 (0.94) | -0.8 (0.94)
Statistical Analysis 1: Comparison: Hyoscine Butylbromide - Tablet vs Hyoscine Butylbromide - Capsule; Test type: Superiority or Other; p = 0.079, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Global Assessment of Efficacy by Patient on 4-point Scale
Description: The endpoint presents global assessment of efficacy: by the patient after 3 days of treatment using a 4-point rating scale (good, satisfactory, not satisfactory, and bad).
Time Frame: Post 3 days of treatment.
Population: Full Analysis Set (FAS): According to the Intent-to-Treat (ITT) principle, all randomized subjects who took at least one dose of study medication and who provided any data for the primary efficacy endpoint were used in FAS.
Measure: Number; unit: Participants
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Number analyzed (Participants) | 143 | 141
Participants
  Good | 35 | 35
  Satisfactory | 69 | 76
  Not satisfactory | 37 | 30
  Bad | 2 | 0

4. Secondary Outcome: Number of Patients With Adverse Events
Description: The endpoint presents number of patients with Adverse Events (AEs). Subjects were required to report spontaneously any AEs as well as the time of onset, end and intensity of these events. Specific questions were asked wherever required or useful to more precisely describe an AE. An Adverse Event was termed serious when one of the following applied: death, directly lifethreatening, continuous or severe impairment, in-patient treatment or prolonging of hospitalization, congenital deformity and other similar medical criteria.
Time Frame: Up to 3 days.
Population: Safety Set (SFS): All randomized subjects who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Number analyzed (Participants) | 146 | 142
Participants
  Subjects with AE | 10 | 10
  Subjects with treatment related AE | 5 | 5
  Subjects with Serious Adverse Event (SAE) | 0 | 0
  AE leading to discontinuation from treatment | 1 | 0
  Subjects with AE: Mild | 10 | 10
  Subjects with AE: Moderate | 0 | 0
  Subjects with AE: Severe | 0 | 0

5. Secondary Outcome: Global Assessment of Tolerability by Investigator on a 4-point Scale
Description: The endpoint presents global assessment of tolerability by subject on a 4-point scale. Global assessment of tolerability regarding all episodes treated by the subject after 3 days of treatment (good, satisfactory, not satisfactory, bad).
Time Frame: Day 3.
Population: Safety Set (SFS): All randomized subjects who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Number analyzed (Participants) | 145 | 141
Participants
  Good | 51 | 47
  Satisfactory | 72 | 72
  Not satisfactory | 21 | 22
  Bad | 1 | 0

6. Secondary Outcome: Number of Subjects With Clinical Relevant Abnormalities for Laboratory, Vital Signs, ElectroCardioGram (ECG) and Physical Examination
Description: Number of patients with findings in clinical relevant abnormalities for laboratory, vital signs, ElectroCardioGram (ECG) and physical examination. Relevant findings or worsening of baseline conditions were reported as Adverse Events (AEs).
Time Frame: Up to 3 days.
Population: Safety Set (SFS): All randomized subjects who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Number analyzed (Participants) | 146 | 142
Participants
  Urinary White Bllood Cell count abnormalities | 4 | 2
  Urinary Red Blood Cell count abnormalities | 2 | 1
  Urinary albumin abnormalities | 1 | 1
  White Blood Cell count abnormalities | 0 | 1
  Platelet count abnormalities | 0 | 1

7. Secondary Outcome: Percentage of Event for Time to Therapeutic Effect
Description: This outcome measure presents percentage of event for time to therapeutic effect defined as the time that the first VAS reduction occurred.
Time Frame: From time of the first dose to the time that the first VAS reduction occurred, up to 180 minutes after the first dose on Day 1.
Population: as for outcome 1
Measure: Number; unit: Percentage of event
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Number analyzed (Participants) | 141 | 140
Percentage of event | 93.6 [NA to NA] | 92.1 [NA to NA]
Statistical Analysis 1: Comparison: Hyoscine Butylbromide - Tablet vs Hyoscine Butylbromide - Capsule; Test type: Superiority or Other; p = 0.531, ANCOVA; Analysis of Covariance (ANCOVA) model including treatment and center as fixed effects and baseline score as covariates was used

ADVERSE EVENTS:
Time Frame: From first drug administration until 3 days after last drug administration, up to 284 days.
Description: The total number of participants at Risk is from SFS [Safety Set] which was different from efficacy set PPS [Per-Protocol Set] and ITT [Intent-to-Treat].
Arm/Group | Hyoscine Butylbromide - Tablet | Hyoscine Butylbromide - Capsule
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/142
Other Adverse Events (participants affected / at risk) | 0/146 | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.